CLINICAL TRIAL: NCT06254820
Title: An Exploratory Study To Establish The Dose, Safety, And Pathogenicity Of A New Influenza B Challenge Strain In Healthy Participants 18 To 55 Years Of Age
Brief Title: Dose, Safety, and Pathogenicity of a New Influenza B Strain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hvivo (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HRD-vCS-002
Record Dates: First submitted 2023-11-14; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Influenza B
Keywords: Influenza; Flu; Human Challenge Trials; Flu B
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: This is an exploratory study of an influenza B challenge strain to determine the optimum infectious titer of challenge agent in healthy participants 18 to 55 years of age
Who Masked: Participant, Investigator
Masking Description: Participant and Investigator. Investigator will be blinded in Part A of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A Dose Arm 1 (Experimental): Medium dose, expected to be approximately 10^6 tissue culture infective dose 50% (TCID50)/mL (titer may be adjusted based on stock titer)
  Interventions: Biological: influenza B/Connecticut/1/21 virus part a dose arm 1
- Part A Dose Arm 2 (Experimental): Dose Arm 2: High dose, expected to be approximately 10^7 TCID50/ mL (titer may be adjusted based on stock titer)
  Interventions: Biological: influenza B/Connecticut/1/21 virus part a dose arm 2
- Part B Dose Extension: (Experimental): Extension of one of the Part A dose arms; which one is to be determined (TBD) depending on outcome of Part A, AND/OR
  Interventions: Biological: influenza B/Connecticut/1/21 virus part b dose 1
- Part B Dose Arm 3 (Experimental): Addition of a 3rd dose, TBD depending on outcome of Part A
  Interventions: Biological: influenza B/Connecticut/1/21 virus part b dose 2

INTERVENTIONS:
Biological: influenza B/Connecticut/1/21 virus part a dose arm 1 — Medium dose, expected to be approximately 10^6 tissue culture infective dose 50% (TCID50)/mL (titer may be adjusted based on stock titer)
  Arms: Part A Dose Arm 1
Biological: influenza B/Connecticut/1/21 virus part a dose arm 2 — High dose, expected to be approximately 10^7 TCID50/ mL (titer may be adjusted based on stock titer)
  Arms: Part A Dose Arm 2
Biological: influenza B/Connecticut/1/21 virus part b dose 1 — Extension of one of the Part A dose arms; which one is to be determined (TBD) depending on outcome of Part A, AND/OR Dose Arm 3
  Arms: Part B Dose Extension:
Biological: influenza B/Connecticut/1/21 virus part b dose 2 — Addition of a 3rd dose, TBD depending on outcome of Part A
  Arms: Part B Dose Arm 3

SUMMARY:
This is an exploratory study of an influenza B challenge strain to determine the optimum infectious titer of challenge agent in healthy participants 18 to 55 years of age.

DETAILED DESCRIPTION:
This is an exploratory study of an influenza B challenge strain to determine the optimum safe infectious titer of challenge agent in healthy participants 18 to 55 years of age. A total of up to 80 participants may be given influenza B challenge virus. The study will be conducted in 2 parts. In Part A, 40 participants will be randomly allocated to one of two groups to be given one of two virus doses (Virus Dose 1 or Virus Dose 2). Based on the outcome of Part A, participants in Part B, may be given Virus Dose 1, Virus Dose 2, or another virus dose (e.g., Virus Dose 3).

Each participant will remain in the study for approximately 1 month from admission to quarantine to the last clinic visit.

The study is divided into three phases:

1. Screening phase: Screening will occur between Day -90 to Day -2/-1. has been signed by the participant.
2. Quarantine phase: Participants will stay in the quarantine unit for approximately 11 days (from Day -2/-1 to Day 8).

   One or two days prior to the day of inoculation with the challenge virus, participants will be admitted to quarantine where their eligibility will be reassessed. If participants remain eligible for the study, they will receive the challenge virus on Day 0. Participants will undergo a range of clinical assessments and safety monitoring for the entirety of their stay in quarantine. Participants will be discharged from the quarantine unit on Day 8 (or may remain longer at the principal investigator's discretion).
3. Outpatient phase: Final follow-up visit 28 days (±3 days) after the day they receive the virus. Their symptoms will be reassessed, and a complete safety examination performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult male or female aged between 18 and 55 years
* A total body weight ≥50 kg and body mass index (BMI) ≥18 kg/m2 and ≤35kg/m2
* In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety.
* Documented medical history
* Adherence to contraception requirements
* Serosuitable for the challenge virus.

Exclusion Criteria:

* History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract (LRT) infection within 4 weeks prior to the first study visit.
* Any history or evidence of any clinically significant or currently active disease.
* Any participants who have smoked ≥10 pack years at any time.
* Female participants who are breastfeeding, or have been pregnant within 6 months prior to the study, or have a positive pregnancy test at any point during screening or prior to inoculation.
* Lifetime history of anaphylaxis and/or a lifetime history of severe allergic reaction.
* Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
* Significant abnormality of the nose, epistaxis, nasal or sinus surgery.
* Recent vaccinations or intention to receive vaccination before the final follow up visit.
* Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned inoculation or planned during the 3 months after the final visit.
* Recent receipt of investigational drugs or challenge viruses.
* Use or anticipated use during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows.
* Positive drugs of abuse test or recent history or presence of alcohol addiction
* A forced expiratory volume in 1 second (FEV1) <80%.
* Positive HIV, hepatitis B virus, or hepatitis C virus test.
* Presence of fever, defined as participant presenting with a temperature reading of ≥37.9C on Day -2/-1 and/or pre-inoculation on Day 0.
* Those employed or immediate relatives of those employed at hVIVO or the sponsor.
* Any other reason, in the opinion of the investigator deems the participant unsuitable for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2024-02-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of AEs and SAEs | Day 0 - Day 28
  Measuring the occurrence of AEs and SAEs as assessed by CTCAE v4.0 during the first 28 days of treatment in >/=40% of participants with laboratory confirmed infection.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Parker, MBBS, Principal Investigator — hVIVO Services Ltd.
Locations (1):
- QMB, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No